CLINICAL TRIAL: NCT06248502
Title: Examining the Relationship Between Pain, Upper Extremity Functionality and Depression in Individuals With Chronic Shoulder Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GaziosmanpasaU_Erol_11
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to examine the relationship between pain, upper extremity functionality and depression in individuals with chronic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Have been suffering from shoulder pain for more than three months

Exclusion Criteria:

* People who have had shoulder surgery

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Shoulder pain
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2024-02-02 (Estimated); Primary Completion 2024-03-02 (Estimated); Study Completion 2024-04-02 (Estimated)

PRIMARY OUTCOMES:
QuickDASH | Baseline
  The level of disability of the patients arising from the upper extremity is determined by evaluating 11 different daily living activities.
Pain Quality Rating Scale | Baseline
  Grading on the scale is between "0" and "10"
Beck Depression Inventory | Baseline
  There are 21 questions with four options for each.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)